CLINICAL TRIAL: NCT03100019
Title: The Effects of Acute Trans-resveratrol Supplementation on Aspects of Cognitive Function and Cerebral Blood Flow, During Hypoxia and Normoxia, in Healthy, Young Humans.
Brief Title: Supplementation of 500mg Trans-resveratrol Within Hypoxic and Normoxic Conditions, in Healthy Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Tim Eschle, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22AX1
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hypoxia, Brain
Keywords: Resveratrol; Cerebral blood flow; Cognition
MeSH Terms: conditions — Hypoxia, Brain | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resveratrol Hypoxia (Experimental): 500mg of trans-resveratrol, tested at a 16% atmospheric oxygen level; the equivalent to 2134m above sea level.
  Interventions: Dietary Supplement: Resveratrol
- Placebo Hypoxia (Placebo Comparator): Pharmaceutical grade fumed silica, tested at a 16% atmospheric oxygen level; the equivalent to 2134m above sea level.
  Interventions: Drug: Placebo
- Resveratrol Normoxia (Experimental): 500mg of trans-resveratrol, tested at a 20.9% atmospheric oxygen level; the equivalent to sea level.
  Interventions: Dietary Supplement: Resveratrol
- Placebo Normoixa (Placebo Comparator): Pharmaceutical grade fumed silica, tested at a 20.9% atmospheric oxygen level; the equivalent to sea level.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol
  Arms: Resveratrol Hypoxia; Resveratrol Normoxia
Drug: Placebo
  Arms: Placebo Hypoxia; Placebo Normoixa

SUMMARY:
Objectives: Resveratrol, a non-flavonoid polyphenol, has been found to consistently modulate cerebral blood flow (CBF) following oral supplementation. Although, this has not resulted in subsequent predicted benefits to cognitive performance in young healthy populations. However, it is argued that those who suffer a reduction in CBF and cognition, such as aging populations, may benefit more from resveratrol administration.

Hypothesis: The current investigation aimed to employ a mild hypoxia as an experimental model of aging in a young healthy population, to assess if resveratrol can attenuate the deficits elicited by the reduction in oxygen supply. It was hypothesized resveratrol would module CBF, to provide a more efficient supply of oxygen to overcome any associated decreases to performance caused by the hypoxic model.

Design: This repeated measures, double blind, placebo controlled, balanced design assessed the cognitive and CBF effects of resveratrol in hypoxia (equivalent to ~2000m above sea level) and normoxia (sea level).

Methods: 24 participants arrived fully fasted (except water) for 12 hrs before completing a baseline measure of a cognitive task battery, and taking the treatment for the day. Following a 45 min absorption period, participants completed 3 full repetitions of the cognitive test battery and, if appropriate, the oxygen level was altered. Changes in CBF were measured by near-infrared spectroscopy throughout the full testing session.

ELIGIBILITY:
Inclusion Criteria:

* Participants who gave informed consent.
* Those who didn't meet any of the exclusion criteria.
* Those who took hormonal contraception (e.g.: the pill, coil, implant, etc.) were allow to participate in the current study.

Exclusion Criteria:

* Smokers.
* People below 18 or above 35 years old at the time of giving consent
* People with Body Mass Index outside of the range 18-35 kg/m2.
* People with blood pressure greater than 140/90 HH/mg
* People who have been living (for more than 3 months) at an altitude of 2000 m or over within the past 6 months.
* People with a history of neurological, vascular or psychiatric illness (excluding depressive illness and anxiety).
* People with a current diagnosis of depression and/or anxiety.
* Participants with learning difficulties, dyslexia or colour blindness.
* Participants with visual impairment that cannot be corrected with glasses or contact lenses.
* Participants with frequent migraines that require medication (more than or equal to 1 per month).
* Participants with disorders of the blood.
* Participants with a heart disorder.
* Participants with a respiratory disorder that requires regular medication (Note: asthma sufferers who only take their medication occasionally/as required are eligible for this study).
* Participants with diabetes.
* Participants with any food intolerances/sensitivities.
* Women who are pregnant, or seeking to become pregnant, or are currently lactating.
* Participants currently taking any prescription medications.
* Participants who have habitually used dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total).
* Participants with a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g., iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation.
* Participants with any health condition that would prevent fulfilment of the study requirements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 2 hours
  Cerebral heamodynamic response (of the prefrontal cortex) at rest and during task performance (all concentration change (μmol / L)).
  There are 3 outputs to this (oxygenated, de-oxygenated and total heamoglobin, detailing changes of oxygenation and de-oxygenation in the neural tissue at rest and during task performance.
Cognitive performance | 1 hour
  Participants completed a number of tasks to measure cognitive domain performance (Episodic Memory, Speed of Attention, & Accuracy of Attention), as part of a 15 minute cognitive battery. Outcomes were measured in accuracy of responses to each task (% correct), reaction time to respond to each task (in milliseconds (ms), and the number of error responses when completing each task.

IPD SHARING:
Plan to Share IPD: No